CLINICAL TRIAL: NCT00486278
Title: A Multi-centre, Randomised, Double-blinded, Controlled, Dose-escalation Trial on Safety and Efficacy of Activated Recombinant FVII Analogue (NN1731) in the Treatment of Joint Bleeds in Congenital Haemophilia Patients With Inhibitors
Brief Title: Haemophilia Patients With Inhibitors Being Treated for Acute Joint Bleeds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1731-1804; 2006-004879-35 (EudraCT Number); CTI-080612 (Other: JAPIC)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2014-12-25 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VII; vatreptacog alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- vatreptacog alfa 5 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)
- vatreptacog alfa 10 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)
- vatreptacog alfa 20 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)
- vatreptacog alfa 40 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)
- vatreptacog alfa 80 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated)
- rFVIIa 90 mcg/kg (Experimental)
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — 90 mcg/kg, injected i.v.
  Arms: rFVIIa 90 mcg/kg
Drug: vatreptacog alfa (activated) — 5 mcg/kg, injected i.v.
  Arms: vatreptacog alfa 5 mcg/kg
Drug: vatreptacog alfa (activated) — 10 mcg/kg, injected i.v.
  Arms: vatreptacog alfa 10 mcg/kg
Drug: vatreptacog alfa (activated) — 20 mcg/kg, injected i.v.
  Arms: vatreptacog alfa 20 mcg/kg
Drug: vatreptacog alfa (activated) — 40 mcg/kg, injected i.v.
  Arms: vatreptacog alfa 40 mcg/kg
Drug: vatreptacog alfa (activated) — 80 mcg/kg, injected i.v.
  Arms: vatreptacog alfa 80 mcg/kg

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Japan, and North and South America.

The aim of this trial is to evaluate the safety and efficacy of activated recombinant human factor VII analogue (vatreptocog alfa (activated)) in haemophilia patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older (at least 18 years in Croatia, France and United Kingdom (UK))
* Clinical diagnosis of congenital haemophilia A or B with a current positive inhibitor titre and a known peak inhibitor of above 5 Bethesda units (BU) (present or in the past) to human FVIII or IX and known antihuman FVIII or IX anamnestic response
* Minimum of 2 joint bleeds (haemarthroses of ankles, knees, or elbows) requiring haemostatic drug treatment within the previous 6 months, or at least 4 joint bleeds (hemarthroses of ankles, knees, or elbows) requiring haemostatic drug treatment within the previous 12 months at trial entry

Exclusion Criteria:

* Known allergy to rFVIIa, and/or suspected allergy to trial product
* Platelet count lower than 50,000 mm^3 based on medical records at trial entry (visit 1)
* Any clinical signs or history of thromboembolic events
* Advanced atherosclerotic disease
* Severe liver disease based on medical records within the past 12 months at trial entry (Visit 1), as defined by alanine aminotransferase (ALAT) above 3 times the upper limit of normal reference range
* Known active pseudo tumours (documented bleeding requiring treatment within the last 3 months
* Subject had any (major) surgical procedure in the 30 days prior to screening into the trial. a. Catheter, ports and dental extractions do not count as surgeries and will not exclude the subject

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (45):
- United States (12):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
- Novo Nordisk Investigational Site, Ciudad Autónoma de Bs. As., Argentina
- Brazil (3):
  - Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, São Paulo
- Novo Nordisk Investigational Site, Edmonton, Alberta, Canada
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Lyon, France
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (3):
  - Novo Nordisk Investigational Site, Castelfranco Veneto
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (5):
  - Novo Nordisk Investigational Site, Hiroshima-shi, Hiroshima
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Warsaw, Poland
- South Africa (3):
  - Novo Nordisk Investigational Site, Parktown Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town
- Novo Nordisk Investigational Site, Madrid, Spain
- Taiwan (2):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Taipei
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] de Paula EV, Kavakli K, Mahlangu J, Ayob Y, Lentz SR, Morfini M, Nemes L, Salek SZ, Shima M, Windyga J, Ehrenforth S, Chuansumrit A; 1804 (adept(TM)1) Investigators. Recombinant factor VIIa analog (vatreptacog alfa [activated]) for treatment of joint bleeds in hemophilia patients with inhibitors: a randomized controlled trial. J Thromb Haemost. 2012 Jan;10(1):81-9. doi: 10.1111/j.1538-7836.2011.04549.x. PMID 22470921
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 sites were initiated globally in 18 countries, including Argentina, Brazil, Canada, Croatia, France, Hungary, Israel, Italy, Japan, Malaysia, Poland, South Africa, Spain, Turkey, Taiwan, Thailand, the United Kingdom and the United States
Pre-assignment Details: A subject could be included in more than one dose escalation cohort with up to one bleeding per cohort, randomised by 4:1 to receive either vatreptacog alfa or rFVIIa 90 (mcg/kg) in a blinded manner.
Groups:
- All Subjects: A total of 51 subjects with 96 qualifying bleeds were treated in the study. A subject could contribute with up to one qualifying bleeding episode per study arm.
Period: Overall Study
Arm/Group | All Subjects
Started | 51 (96 bleeds by 51 subjects, 77 were treated with vatreptacog alfa and 19 with rFVIIa)
Completed | 42
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs)
Description: Adverse event is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Monitoring of adverse events was performed from start of the trial to approximately 4 weeks after administration of trial product.
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: events
Groups:
- Vatreptacog Alfa 5 mcg/kg: Subjects received vatreptacog alfa 5 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to one qualifying bleeding episode per vatreptacog alfa arm.
- Vatreptacog Alfa 10 mcg/kg: Subjects received vatreptacog alfa 10 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to one qualifying bleeding episode per vatreptacog alfa arm.
- Vatreptacog Alfa 20 mcg/kg: Subjects received vatreptacog alfa 20 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to one qualifying bleeding episode per vatreptacog alfa arm.
- Vatreptacog Alfa 40 mcg/kg: Subjects received vatreptacog alfa 40 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to one qualifying bleeding episode per vatreptacog alfa arm.
- Vatreptacog Alfa 80 mcg/kg: Subjects received vatreptacog alfa 80 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to one qualifying bleeding episode per vatreptacog alfa arm.
- rFVIIa 90 mcg/kg: Subjects received rFVIIa standard dose regimen 90 mcg/kg intravenously every 3 hours (+ 30 minutes) maximum of 3 times until bleeding was controlled. A subject could contribute with up to 5 qualifying bleeding episode per to the rFVIIa arm, corresponding to number of dose escalation cohorts.
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
events
  All AEs | 10 | 8 | 5 | 5 | 0 | 11
  Serious AEs | 3 | 5 | 2 | 2 | 0 | 3

2. Secondary Outcome: Activated Recombinant Human Factor VII Analogue Activity in the Blood
Time Frame: 0-24 hours after trial product administration
Population: All randomised patients in top three dosing tiers 3, 4 and 5 who had pharmacokinetic assessments and completed the trial without violation of the protocol in a manner that was judged to affect the pharmacokinetic endpoints were included in the pharmacokinetic analysis set.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 16 | 16 | 10 | 17
IU/mL
  Pre-dose |  |  | 0.1 (0.1) | 0.1 (0) | 0 (0) | 0.1 (0)
  1 hours post-dose |  |  | 5.3 (1.3) | 12.8 (5.3) | 19.7 (7.2) | 28.0 (12.6)
  12 hours post-dose |  |  | 0.4 (0.4) | 2.3 (4.5) | 0.3 (0.3) | 14.1 (27.3)
  24 hours post-dose |  |  | 0 (0) | 0 (0) | 0 (0) | 0.1 (0)

3. Secondary Outcome: Prothrombin Time (PT)
Description: The test measures the clotting time of plasma following the activation of tissue factor (TF also called thromboplastin) and calcium to hypocalcemic plasma. PT was provided in percent based on the measured PT in seconds and related/converted with the relevant standard curve. The percent value was derived based on the hyperbolic relation between PT (sec) and % PT activity.
Time Frame: pre-dose - 12 hours after trial product administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
percentage (%)
  Pre-dose | 80.1 (12.6) | 77.6 (19.1) | 79.1 (14.9) | 85.9 (15.5) | 85.5 (8.8) | 88.3 (25.6)
  1 hours post-dose | 84.3 (16.3) | 99.6 (17.9) | 112.1 (14.6) | 123.4 (14.7) | 128.5 (7.6) | 139.0 (0)
  12 hours post-dose | 82.1 (16.2) | 73.2 (19.2) | 86.9 (14.1) | 94.5 (17.5) | 92.3 (16.8) | 112.1 (29.1)

4. Secondary Outcome: F1 + 2 (Prothrombin Fragments 1+2)
Description: Thrombin and F1+2 are formed in equimolar quantities by the enzymatic cleavage of prothrombin (FII), and F1+2 thus indicate that thrombin has been generated.
Time Frame: pre-dose - 12 hours after trial product administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
pmol/L
  Pre-dose | 289.8 (310.9) | 131.8 (48.7) | 139.1 (50.4) | 121.2 (34.5) | 125.4 (45.9) | 169.3 (56.9)
  1 hour post-dose | 443.7 (414.7) | 241.7 (162.0) | 401.6 (292.6) | 365.9 (145.4) | 385.7 (88.8) | 309.7 (284.5)
  12 hour post-dose | 325.9 (299.4) | 198.9 (250.9) | 158.6 (54.5) | 199.8 (91.5) | 136.9 (43.8) | 268.2 (158.0)

5. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT)
Description: The aPTT time measured in clinical samples reflects both the effect of the drugs (generation of thrombin and FXa) and the presence of rFVIIa /rFVIIa analogue in the plasma samples causing a dose dependent shortening of the clotting time.
Time Frame: pre-dose - 12 hours after trial product administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sec
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
Sec
  Pre-dose | 120.6 (22.6) | 126.0 (26.4) | 122.8 (15.9) | 119.2 (31.3) | 117.4 (17.9) | 113.8 (17.4)
  1 hours post-dose | 102.1 (19.4) | 79.7 (13.9) | 68.7 (15.7) | 52.8 (14.1) | 48.6 (24.0) | 70.0 (9.8)
  12 hours post-dose | 111.7 (22.4) | 107.9 (27.7) | 107.9 (14.8) | 104.4 (31.2) | 99.3 (19.6) | 98.6 (20.8)

6. Secondary Outcome: Cessation of Bleeding: Number of Doses Needed to Control Bleeding
Time Frame: Within 9 hours after first trial product administration or need of additional haemostatic medication within 9 hours after first trial administration additional haemostatic agents required to control bleed (treatment failure)
Population: All randomised patients for whom at least one of the efficacy variables is assessed were to be included in the full analysis set (FAS). For the outcome measure 1 subject did not contribute to the data.
Measure: Number; unit: bleeding episodes
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 15 | 19 | 16 | 16 | 10 | 17
bleeding episodes
  1 dose | 3 | 3 | 2 | 5 | 4 | 6
  2 doses | 5 | 9 | 7 | 6 | 4 | 4
  3 doses | 4 | 4 | 7 | 4 | 2 | 7
  treatment failure | 3 | 3 | 0 | 1 | 0 | 2

7. Secondary Outcome: Number of Subjects With Need for Additional Haemostatic Agents
Time Frame: within 24 hours after successful control of bleeding episode with trial product
Population: All randomised patients for whom at least one of the efficacy variables is assessed were to be included in the full analysis set (FAS). For the outcome measure 9 subjects did not contribute to the data.
Measure: Number; unit: participants
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 12 | 16 | 16 | 15 | 10 | 17
participants | 4 | 1 | 1 | 1 | 1 | 1

8. Secondary Outcome: Pharmacokinetic Parameters Based on FVIIa Activity: AUC 0-t (Area Under the Plasma FVIIa Activity-time Curve From Time Zero to the Time (t) )
Time Frame: 0-24 hours after trial product administration
Population: All randomised patients in top 3 dosing tiers 3, 4 and 5 who had pharmacokinetic assessments and completed the trial without violating the protocol in a manner that was judged to affect the pharmacokinetic endpoints were included in the pharmacokinetic analysis set. Some subjects did not contribute for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU*h)/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 7 | 7
(IU*h)/mL |  |  | 34.24 (27.00) | 66.85 (50.51) | 136.19 (18.56) | 74.35 (45.30)

9. Secondary Outcome: Pharmacokinetic Parameters Based on FVIIa Activity: AUC(0-inf) (Area Under the Plasma FVIIa Activity-time Curve From Time Zero to Infinity)
Time Frame: 0-24 hours after trial product administration
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU*h)/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 7 | 7
(IU*h)/mL |  |  | 35.76 (26.34) | 71.23 (55.42) | 139.63 (18.35) | 101.38 (40.77)

10. Secondary Outcome: Pharmacokinetic Parameters Based on FVIIa Activity: MRT (Mean Residence Time)
Time Frame: 0-24 hours after trial product administration
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 7 | 7
hours |  |  | 0.68 (0.16) | 0.88 (0.33) | 0.56 (0.10) | 2.23 (0.54)

11. Secondary Outcome: Pharmacokinetic Parameters Based on FVIIa Activity: t½ (Terminal Half-life)
Time Frame: 0-24 hours after trial product administration
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 13 | 11 | 7 | 7
hours |  |  | 0.92 (0.18) | 1.28 (1.28) | 0.71 (0.16) | 1.66 (0.35)

12. Secondary Outcome: Pharmacokinetic Parameters Based on FVIIa Activity: CL (Total Clearance)
Time Frame: 0-24 hours after trial product administration
Population: as for outcome 8
Measure: Median (Full Range); unit: mL/h
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 7 | 7
mL/h |  |  | 9365.8 [6829.8 to 15065] | 11247 [5315.6 to 21314] | 10409 [6262.9 to 13276] | 3078.3 [1636.9 to 5039.4]

13. Secondary Outcome: Pharmakokinetic Parameters Based on FVIIa Activity: Vss (Distribution Volume at Steady State)
Time Frame: 0-24 hours after trial product administration
Population: as for outcome 8
Measure: Median (Full Range); unit: mL/kg
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 7 | 7
mL/kg |  |  | 5396.9 [3319.1 to 12215] | 9597.0 [5522.7 to 18310] | 5538.7 [4210.7 to 6482.6] | 6696.7 [3037.3 to 10328]

14. Secondary Outcome: Immunogenicity (Inhibitor Development)
Description: Immunogenicity was tested by formation of neutralising antibodies towards vatreptacog alfa and/or rFVIIa.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
participants | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Biochemistry: ALAT (Alanine Aminotransferase)
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
U/L
  Screening | 26.0 (18.7) | 32.8 (31.3) | 30.6 (27.1) | 39.3 (33.3) | 24.2 (17.9) | 30.1 (21.4)
  Pre-dose | 22.7 (19.9) | 29.9 (23.0) | 32.4 (37.1) | 29.1 (16.4) | 28.1 (16.6) | 49.4 (73.7)
  12 hours post-dose | 20.1 (16.8) | 25.6 (19.2) | 21.4 (15.4) | 30.9 (18.2) | 24.5 (14.4) | 45.1 (66.0)

16. Secondary Outcome: Biochemistry: Creatinine
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
micromol/L
  Screening | 66.9 (23.6) | 67.2 (13.8) | 63.6 (23.3) | 67.7 (15.7) | 60.0 (17.3) | 66.9 (16.0)
  Pre-dose | 68.2 (23.3) | 70.1 (10.0) | 69.8 (15.3) | 69.1 (19.1) | 67.7 (10.8) | 71.1 (15.2)
  12 hours post-dose | 58.3 (23.6) | 63.1 (17.7) | 70.6 (16.8) | 71.9 (15.2) | 68.0 (10.7) | 70.6 (14.8)

17. Secondary Outcome: Haematology: Haemoglobin
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
g/dL
  Screening | 13.9 (1.8) | 14.7 (1.6) | 14.2 (1.4) | 14.2 (1.8) | 14.6 (1.3) | 13.8 (1.3)
  Pre-dose | 13.8 (2.3) | 14.6 (1.7) | 14.4 (1.2) | 13.9 (2.1) | 14.8 (1.3) | 14.1 (1.3)
  12 hours post-dose | 13.5 (2.2) | 13.9 (1.7) | 13.7 (1.2) | 13.0 (2.2) | 14.2 (0.8) | 13.5 (1.3)

18. Secondary Outcome: Haematology: Red Cell Count
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
10^12 cells/L
  Screening | 5.0 (0.5) | 5.4 (0.9) | 5.3 (1.0) | 5.1 (0.4) | 5.7 (1.2) | 5.3 (1.0)
  Pre-dose | 5.1 (0.5) | 5.1 (0.4) | 5.2 (0.4) | 5.1 (0.4) | 5.1 (0.4) | 5.2 (0.5)
  12 hours post-dose | 5.0 (0.7) | 4.9 (0.4) | 4.9 (0.3) | 4.8 (0.5) | 4.9 (0.3) | 5.0 (0.6)

19. Secondary Outcome: Haematology: Packed Cell Volume
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
percentage (%)
  Screening | 41.6 (5.1) | 43.7 (3.9) | 42.2 (3.6) | 42.4 (4.3) | 44.0 (3.3) | 41.6 (3.8)
  Pre-dose | 41.3 (6.1) | 43.1 (4.0) | 42.6 (3.2) | 42.5 (6.3) | 44.6 (4.6) | 42.3 (3.5)
  12 hours post-dose | 40.6 (6.0) | 40.9 (4.0) | 40.6 (2.9) | 39.9 (6.8) | 42.2 (2.9) | 40.4 (3.8)

20. Secondary Outcome: Haematology: White Cell Count
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
10^9 cells/L
  Screening | 6.7 (1.9) | 6.3 (2.5) | 7.2 (2.4) | 6.9 (2.7) | 6.6 (1.5) | 5.8 (1.8)
  Pre-dose | 7.6 (2.3) | 7.3 (2.6) | 7.8 (1.9) | 7.1 (2.2) | 7.1 (2.3) | 6.5 (2.1)
  12 hours post-dose | 7.7 (3.4) | 7.2 (2.1) | 8.2 (2.0) | 7.3 (2.6) | 6.8 (1.4) | 7.1 (2.5)

21. Secondary Outcome: Haematology: Platelet Count
Time Frame: screening visit, pre-dose and 12 hours after dosing
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Number analyzed (Participants) | 16 | 19 | 16 | 16 | 10 | 17
10^9 cells/L
  Screening | 259.8 (96.2) | 253.8 (82.9) | 250.8 (61.2) | 276.1 (75.5) | 272.5 (73.2) | 259.0 (86.1)
  Pre-dose | 253.5 (90.5) | 248.6 (65.2) | 252.7 (50.8) | 278.8 (78.0) | 278.1 (59.0) | 271.1 (82.4)
  12 hours post-dose | 242.7 (83.7) | 244.8 (57.4) | 255.8 (61.9) | 287.0 (94.8) | 266.8 (53.1) | 260.7 (69.4)

ADVERSE EVENTS:
Time Frame: Monitoring of adverse events was performed from start of the trial to approximately 4 weeks after administration of trial product.
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product.
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 40 mcg/kg | Vatreptacog Alfa 80 mcg/kg | rFVIIa 90 mcg/kg
Serious Adverse Events (participants affected / at risk) | 2/16 | 3/19 | 2/16 | 2/16 | 0/10 | 2/19
Other Adverse Events (participants affected / at risk) | 6/16 | 3/19 | 3/16 | 1/16 | 0/10 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatreptacog Alfa 5 mcg/kg (N=16) | Vatreptacog Alfa 10 mcg/kg (N=19) | Vatreptacog Alfa 20 mcg/kg (N=16) | Vatreptacog Alfa 40 mcg/kg (N=16) | Vatreptacog Alfa 80 mcg/kg (N=10) | rFVIIa 90 mcg/kg (N=19)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Removal of foreign body from joint (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatreptacog Alfa 5 mcg/kg (N=16) | Vatreptacog Alfa 10 mcg/kg (N=19) | Vatreptacog Alfa 20 mcg/kg (N=16) | Vatreptacog Alfa 40 mcg/kg (N=16) | Vatreptacog Alfa 80 mcg/kg (N=10) | rFVIIa 90 mcg/kg (N=19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Teeth brittle (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained during the conduct of this trial is considered confidential and can be used by Novo Nordisk for regulatory purposes and for the general development of the trial product. The information obtained during this trial may be made available to other physicians who are conducting other clinical trials with the trial product, if deemed necessary by Novo Nordisk.